CLINICAL TRIAL: NCT03860753
Title: Effects of Pioglitazone on Stress Reactivity and Alcohol Craving (Pilot)
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Halted enrollment due to COVID-19
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Jin Ho Yoon, Assistant Professor, The University of Texas Health Science Center, Houston
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HSC-MS-18-0922 (pilot)
Record Dates: First submitted 2019-02-28; First posted 2019-03-04 (Actual); Results first posted 2020-10-26 (Actual); Last update posted 2020-10-26 (Actual); Status verified 2020-10

CONDITIONS: Alcohol Use Disorder
Keywords: Alcohol; Pioglitazone; Stress; Anxiety
MeSH Terms: conditions — Alcoholism; Anxiety Disorders | interventions — Pioglitazone

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Pioglitazone (Experimental)
  Interventions: Drug: Pioglitazone
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Pioglitazone — For the current trial we will follow recommended adult initial dosing at 30 mg/d to reach maintenance dose of 45 mg/d by week 2, which is within standard titration parameters as per the investigator's brochure.
  Arms: Pioglitazone
Drug: Placebo — Pill capsules will look same as that of active drug.
  Arms: Placebo

SUMMARY:
The purpose of this study is to assess the effect of pioglitazone on stress- and alcohol-related measures in treatment-seeking individuals with alcohol use disorder (AUD) and elevated levels of stress and anxiety.

ELIGIBILITY:
Inclusion Criteria:

* treatment-seeking individuals diagnosed with AUD diagnostic statistical manual 5 (DSM-5)
* fluent in English
* past month excessive alcohol use (>7 drinks/week for woman, >14 drinks/week for men, >3 drinks/occasion for women>4 drinks/occasion for men)14
* baseline Hamilton Anxiety Rating Scale (HAM-A) or Perceived Stress Scale (PSS) core indicative of mild to moderate anxiety (score 8 to 23) or moderate stress (score 14 to 26), respectively
* increase in alcohol craving following the baseline stress reactivity assessment.

Exclusion Criteria:

* Individuals will be excluded for exhibiting severe scores on the HAM-A, PSS, or post-traumatic (PTSD) checklist (PCL-5) at the discretion of the admitting physician
* physical dependence on alcohol Alcohol Use Disorders Inventory (AUDIT) score indicative of severe alcohol dependence (≥13 for women, ≥15 for men)
* greater than mild substance use disorder on drugs other than alcohol, nicotine, and marijuana
* contraindications for taking pioglitazone; medical conditions contraindicating pioglitazone pharmacotherapy or taking contraindicated medications
* be pregnant, nursing, or planning on becoming pregnant during the course of the study
* have any other illness, condition, or use of medications, which in the opinion of the PI and/or admitting physician would preclude safe and/or successful completion of the study.

Ages: 21 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 4 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2019-08-23 (Actual); Study Completion 2019-08-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jin H Yoon, PhD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas Health Science at Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Pioglitazone | Placebo
Started | 4 | 0
Completed | 4 | 0
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: All 4 participants were allocated to Pioglitazone and none to placebo.
Groups:
- Total: Total of all reporting groups
Arm/Group | Pioglitazone | Placebo | Total
Number analyzed (Participants) | 4 | 0 | 4
Age, Continuous [Mean (Standard Deviation); unit: years] | 30.5 (5.20) |  | 30.5 (5.20)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 1
  Male | 3 | 0 | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 3 | 0 | 3
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 0 | 2
  White | 2 | 0 | 2
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 4 | 0 | 4

OUTCOME MEASURES:

1. Primary Outcome: Change in Stress-reactivity as Assessed by Heart Rate Change During the Cold Pressor Task (CPT)
Description: The cold pressor task (CPT) a stress-inducer in human laboratory studies that elicits moderate activation of the sympathetic nervous system and limited activation of the HPA-axis. During CPT, participants will submerge their dominant arm in an ice-water bath for up to 2 minutes, and heart rate will be measured before and after CPT. The heart rate change for each time point is calculated as heart rate after CPT minus the heart rate before CPT. This outcome measure reports the heart rate change at week 4 minus the heart rate change at baseline.
Time Frame: baseline, week 4
Population: All 4 participants were allocated to Pioglitazone and none to placebo.
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | Pioglitazone | Placebo
Number analyzed (Participants) | 4 | 0
beats per minute | -4.67 (11.60) |

2. Primary Outcome: Change in Stress-reactivity as Assessed by Change in Systolic Blood Pressure During the Cold Pressor Task (CPT)
Description: The cold pressor task (CPT) a stress-inducer in human laboratory studies that elicits moderate activation of the sympathetic nervous system and limited activation of the HPA-axis. During CPT, participants will submerge their dominant arm in an ice-water bath for up to 2 minutes, and blood pressure will be measured before and after CPT. The blood pressure change for each time point is calculated as blood pressure after CPT minus the blood pressure before CPT. This outcome measure reports the blood pressure change at week 4 minus the blood pressure change at baseline.
Time Frame: baseline, week 4
Population: All 4 participants were allocated to Pioglitazone and none to placebo.
Measure: Mean (Standard Deviation); unit: millimeters of mercury (mmHg)
Arm/Group | Pioglitazone | Placebo
Number analyzed (Participants) | 4 | 0
millimeters of mercury (mmHg) | -2.67 (0.58) |

3. Primary Outcome: Change in Stress-reactivity as Assessed by Diastolic Blood Pressure Change During the Cold Pressor Task (CPT)
Description: as for outcome 2
Time Frame: baseline, week 4
Population: All 4 participants were allocated to Pioglitazone and none to placebo.
Measure: Mean (Standard Deviation); unit: millimeters of mercury (mmHg)
Arm/Group | Pioglitazone | Placebo
Number analyzed (Participants) | 4 | 0
millimeters of mercury (mmHg) | -7.67 (8.08) |

4. Primary Outcome: Change in Stress-reactivity as Assessed by Salivary Cortisol Level Change During the Cold Pressor Task (CPT)
Description: The cold pressor task (CPT) a stress-inducer in human laboratory studies that elicits moderate activation of the sympathetic nervous system and limited activation of the HPA-axis. During CPT, participants will submerge their dominant arm in an ice-water bath for up to 2 minutes, and salivary cortisol level will be measured before and after CPT. The salivary cortisol level change for each time point is calculated as salivary cortisol level after CPT minus the salivary cortisol level before CPT. This outcome measure reports the salivary cortisol level change at week 4 minus the salivary cortisol level change at baseline.
Time Frame: baseline, week 4
Population: All 4 participants were allocated to Pioglitazone and none to placebo.
Measure: Mean (Standard Deviation); unit: picograms per milliliter (pg/mL)
Arm/Group | Pioglitazone | Placebo
Number analyzed (Participants) | 4 | 0
picograms per milliliter (pg/mL) | -108.07 (830.46) |

5. Primary Outcome: Change in Stress-reactivity as Assessed by Self-report on a Visual Analogue Scale (VAS)
Description: The visual analogue scale (VAS) ranges from 0-10, with a higher score indicating higher stress.
Time Frame: baseline, week 4
Population: All 4 participants were allocated to Pioglitazone and none to placebo.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Pioglitazone | Placebo
Number analyzed (Participants) | 4 | 0
units on a scale | -1.33 (1.53) |

6. Secondary Outcome: Change in Alcohol Use as Indicated by Self Report Using the Alcohol Timeline Followback (TLFB)
Description: The Alcohol Timeline Followback (TLFB) is a drinking assessment method that obtains an estimate of daily drinking. Participants provide a retrospective estimate of the number of drinks per week for the last seven days.
Time Frame: baseline, week 4
Population: All 4 participants were allocated to Pioglitazone and none to placebo.
Measure: Mean (Standard Deviation); unit: number of drinks per week
Arm/Group | Pioglitazone | Placebo
Number analyzed (Participants) | 4 | 0
number of drinks per week | -13.38 (11.22) |

7. Secondary Outcome: Change in Alcohol Craving as Assessed by Self Report Using the The Penn Alcohol Craving Scale (PACS).
Description: The Penn Alcohol Craving Scale (PACS) is a 5-item questionnaire that measures an individual's craving to drink alcohol in the past week. Each item is scored on a scale from 0 to 6, with a total score range of 0 to 30. A higher score indicates greater level of alcohol craving.
Time Frame: baseline, week 4
Population: All 4 participants were allocated to Pioglitazone and none to placebo.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Pioglitazone | Placebo
Number analyzed (Participants) | 4 | 0
score on a scale | -8.5 (6.6) |

ADVERSE EVENTS:
Time Frame: 4 weeks
Description: All 4 participants were allocated to Pioglitazone and none to placebo.
Arm/Group | Pioglitazone | Placebo
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/0
Other Adverse Events (participants affected / at risk) | 2/4 | 0/0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pioglitazone (N=4) | Placebo (N=0)
weight gain (General disorders) | 2 (2) | 0 (0)
right ankle stiffness (General disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
Early termination leading to small numbers of subjects analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-05-08): https://cdn.clinicaltrials.gov/large-docs/53/NCT03860753/Prot_SAP_000.pdf